CLINICAL TRIAL: NCT01695057
Title: A Pilot Clinical Trial to Evaluate the Biological Activity of HDAC (Histone Deacetylase Transferases) Inhibition on ER and PR Expression in Triple Negative Invasive Breast Cancer
Brief Title: Vorinostat Before Surgery in Treating Patients With Triple-Negative Breast Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1B-10-10; NCI-2012-01612 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Stage II Breast Cancer; Stage IIIA Breast Cancer; Triple-negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (vorinostat and surgery) (Experimental): Patients receive vorinostat 400 mg daily PO on days 1-21 followed by surgery within 14 days.
  Interventions: Drug: vorinostat; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: vorinostat — Given PO
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Procedure: therapeutic conventional surgery — Undergo surgery
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies vorinostat before surgery in treating patients with triple-negative breast cancer. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving enzyme inhibitor therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the ability of histone deacetylase (HDAC) inhibition using suberoylanilide hydroxamic acid (SAHA) (vorinostat) to induce expression of the estrogen receptor (ER) and progesterone receptor (PR) genes in solid human triple negative invasive breast cancer.

OUTLINE:

Patients receive vorinostat 400 mg daily orally (PO) on days 1-21 followed by surgery within 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Resectable tumor measuring 2cm or more
* Histologically documented, newly diagnosed, triple negative invasive breast cancer characterized by 0% immunohistochemistry (IHC) nuclear staining for ER-alpha, 0% IHC nuclear staining for PR-alpha, and no amplification of human epidermal growth factor receptor 2 (HER2)/neu by fluorescent in situ hybridization (FISH) using institutional standard; standard IHC assays for ER and PR use antibodies to ER-alpha and PR-alpha and PR-beta
* Southwest Oncology Group (SWOG) performance status of less than or equal to 1
* Absolute neutrophil count (ANC) >= 1500/uL
* Hemoglobin (Hgb) >= 9 g/dL
* Platelets >= 100,000/uL
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamic pyruvate transaminase (SGPT) =< 2.5 x upper limit of normal (ULN) or =< 5.0 x ULN in patients with liver metastases
* Creatinine =< 2.0 mg/dL or calculated creatinine clearance >= 50 ml/min
* Albumin >= 3 g/dL
* Potassium >= lower limit normal (LLN)
* Phosphorous >= LLN
* Calcium >= LLN
* Magnesium > LLN
* Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to start of treatment
* Accessible for treatment and follow-up
* Written informed consent prior to study entry

Exclusion Criteria:

* HER2/neu amplification by FISH
* Concurrent neoadjuvant anti-cancer treatment with chemotherapy, endocrine therapy, biologically targeted therapy or radiotherapy
* Known hypersensitivity to SAHA
* Preexisting hepatic impairment or renal impairment
* Intent to receive additional neoadjuvant therapy prior to surgery
* Concurrent use of an HDAC inhibitor or hydralazine
* Known diagnosis of human immunodeficiency virus (HIV) infection
* Major surgery < 4 weeks prior to starting study drug
* Pregnant or breastfeeding or female of reproductive potential not using an effective method of birth control
* Other concurrent severe, uncontrolled infection or intercurrent illness, including but not limited to ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
* Prior antiestrogens (selective estrogen receptor modulator [SERM] or aromatase inhibitors) within 6 months of study entry
* Underlying medical, psychiatric or social conditions that would preclude patient from receiving treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2014-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Combined PR/ER response | 21 days
  The proportion of patients who achieve sufficient deacetylation of ER and PR will be estimable with a standard error no greater than +/- 0.05. The proportion of patients who exhibit a sufficient change in ER or PR expression can be estimated with similar precision. In addition, paired t-tests and McNamaraÃ¢s test will be used to evaluate whether the effect of vorinostat on deacetylation status or gene expression differs between ER or PR, and linear regression analysis will be used to evaluate the association between deacetylation changes and corresponding expression changes in ER and PR genes.

SECONDARY OUTCOMES:
Grade 3 or 4 toxicities using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Within 3 days prior to surgery
  The toxicities observed will be summarized in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity (by NCI Common Toxicity Criteria v4.0 and nadir or maximum values for the laboratory measures), time of onset (i.e. week of treatment), duration, and reversibility or outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Agustin Garcia, Principal Investigator — University of Southern California